CLINICAL TRIAL: NCT06643910
Title: A Study on the Safety and Efficacy of BST08 in Treating Advanced Non-Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BioSyngen Pte Ltd (Industry)
Collaborators: South China Hospital of Shenzhen University (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BR-BST08-001
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BST08 (Experimental): Intravenous infusion
  Interventions: Biological: Single drug group A; Biological: Combined treatment group B

INTERVENTIONS:
Biological: Single drug group A — 9x10^10 BST08 cells, Intravenous infusion，3 subject is planned to be enrolled
Biological: Combined treatment group B — 9x10^10 BST08 cells+ Pembrolizumab Injection，200mg，Q3W, Intravenous infusion，6subject is planned to be enrolled

SUMMARY:
This study is an exploratory clinical trial initiated by an open, single arm researcher to evaluate the safety, tolerability, and preliminary efficacy of BST08 in the treatment of advanced non-small cell lung cancer in subjects. This study plans to set up two experimental groups: monotherapy group A: 9x10 ^ 10 BST08 (3 cases) and combination therapy group B: 9x10 ^ 10 BST08+Pabolizhu 200mg Q3W (6 cases).

DETAILED DESCRIPTION:
Main purpose:

Evaluate the safety and tolerability of BST08 treatment in subjects with advanced non-small cell lung cancer.

Secondary purpose:

1. Evaluate the preliminary effectiveness of BST08 in the treatment of advanced non-small cell lung cancer subjects;
2. Evaluate the pharmacokinetic (PK) characteristics of BST08.

ELIGIBILITY:
Inclusion Criteria:

* 1: Age 18-70 years old (including the critical value);
* 2: Non-small cell lung cancer diagnosed by histopathology or cytology without driver mutation progresses after receiving at least second-line systemic therapy including anti-PD-1 /L1 monoclonal antibody.
* 3: At least one tumor lesion has not received radiation therapy or other local treatment within 28 days. In addition, according to the researchers' judgment, at least 2 tumor puncture samples (from different lesions) with good integrity and ≥2cm length can be obtained by surgical resection or puncture for the preparation of BST08.
* 4: At least one measurable lesion as defined by the RECIST 1.1 standard;
* 5: Eastern Cooperative Oncology Group (ECOG) score ≤1 score;
* 6: Expected survival time ≥3 months;
* 7: Adequate organ and bone marrow function during the screening and preparation phase (within 14 days prior to tumor tissue sampling)
* 8: Prior to the tumor tissue sampling, the adverse reactions caused by previous treatment had returned to the Common Adverse Event Evaluation Criteria (CTCAE) 5.0≤2 (except for alopecia, peripheral neurotoxicity of grade 2 or below, and other toxicities that researchers judged to have no safety risk);
* 9: From the signing of the informed consent to the acceptance of effective contraceptive measures within 6 months after the BST08 infusion (subjects must use non-drug contraceptive measures);
* 10: Those who fully understand the test and voluntarily sign the informed consent, and can comply with the visit and related procedures stipulated in the program

Exclusion Criteria:

* 1: Pregnant or lactating women;
* 2. Subjects with a history of severe allergy to the experimental drug, including but not limited to cyclophosphamide, fludarabine, and BST08 components;
* 3: Past or current presence of hepatic encephalopathy; Other patients with known uncontrolled or untreated central nervous system metastases; Patients with stable symptoms who had received treatment and stopped treatment with corticosteroids and anticonvulsants ≥4 weeks prior to preconditioning were excluded;
* 4: Extensive liver metastasis was confirmed (imaging estimated tumor volume accounted for ≥50% of the total liver volume);
* 5: Organ transplantation, hematopoietic stem cell transplantation history;
* 6. Other serious medical conditions that may limit participants' participation in this trial
* 7: HIV positive, or treponema pallidum antibody positive;
* 8: Active hepatitis B infection, defined as Hepatitis B core antibody (HBcAb) or Hepatitis B surface antigen (HBsAg) positive with HBV-DNA> 10,000 IU/ml, or 200 IU. Or hepatitis C, defined as HCV RNA above the lower limit for clinical trial center detection. These patients will need to continue taking antiviral drugs during the study period;
* 9: Any immunosuppressive drugs, such as corticosteroids, were used in the 4 weeks prior to the tumor tissue sampling, or co-existing diseases were determined by the investigator to require the use of immunosuppressive drugs during the trial. However, the use of physiological doses of corticosteroids (i.e., no more than 15mg/ day of prednisone or equivalent doses of other corticosteroids) is permitted, and the use of corticosteroids for inhalation, intranasal, topical or prophylactic use of contrast media allergies is permitted;
* 10: Local treatment such as interventional therapy, radiotherapy, ablation and systemic treatment (including small molecule targeted drugs, anti-PD-1 / PD-L1 monoclonal antibodies and chemotherapy, etc.) had been received within 4 weeks before pretreatment. Or received thymosin, interferon and other immunotherapy or any Chinese herbal medicine or proprietary Chinese medicine for tumor control within 1 week prior to pretreatment;
* 11: Those who have received live vaccine within 3 months prior to screening or plan to receive live vaccine during the trial;
* 12: Patients who underwent major surgery (≥ Grade 3 surgery) within 4 weeks prior to screening, or who required elective surgery during the trial period (other than tumor tissue sampling surgery/puncture);
* 13: Patients who had surgical complications or delayed wound healing prior to pretreatment, and who were judged by the investigators to increase the risk of eluviation, TIL treatment, or infection;

  14: diagnosed with other primary malignancies within 5 years prior to screening, excluding radical basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and/or radical resection of carcinoma in situ;
* 15: Genetically modified cell therapy products received 6 months before pretreatment;
* 16: Participants with known alcohol, drug, or substance abuse and other conditions deemed inappropriate by the researchers to participate in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-10-24 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) | From the infusion (Day 0) to Day 28
  DLT is defined as the following adverse events related to the investigational drug (definitely related, likely related, possibly related) that occur within 28 days after administration of BST08 (using CTCAE 5.0 or CRS grading criteria): (1) hematological toxicity; (2) Grade 3 non hematological toxicity lasting for more than 7 days, or ≥ Grade 4 non hematological toxicity, regardless of duration, but excluding the following situations; (3)Cytokine Release Syndrome(CRS)
Maximum ToleratedDose（MTD） | From the infusion (Day 0) to Day 28
  The highest dose of DLT observed in subjects with less than 2/6 (at least 6 subjects in this experimental group received BST08 administration and completed DLT observation)

CONTACTS AND LOCATIONS:
Overall Officials: Yuqing Li, PhD, Principal Investigator — South China Hospital of Shenzhen University; Mingyong Han, PhD, Principal Investigator — South China Hospital of Shenzhen University
Locations (1):
- Yuqing Li, Shenzhen, Guangdong, China